CLINICAL TRIAL: NCT03053570
Title: Study Comparing Pulmonary Vein Isolation With the Cryoballoon and Radiofrequency Energy(Contact Force) in the Treatment of Persistent Atrial Fibrillation (PerAF)
Brief Title: Study Comparing Pulmonary Vein Isolation With the Cryoballoon and Radiofrequency Energy(Contact Force) in the Treatment of Persistent Atrial Fibrillation (AF) (Cryo Vs CF in PerAF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Cardiometabolic Registries (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cryo Vs CF in PerAF
Record Dates: First submitted 2017-01-31; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Cryoballoon; Contact Force; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon (Experimental)
  Interventions: Device: Cryoballoon; Device: Radiofrequency Energy(Contact Force)
- Radiofrequency Energy(Contact Force) (Experimental)
  Interventions: Device: Cryoballoon; Device: Radiofrequency Energy(Contact Force)

INTERVENTIONS:
Device: Cryoballoon — use Cryoballoon to isolation the Pulmonary Vein
Device: Radiofrequency Energy(Contact Force) — use Radiofrequency Energy(Contact Force) to isolation the Pulmonary Vein

SUMMARY:
The purpose of this study is to perform a prospective, randomised study investigating the safety and efficacy of cryoballoon catheter ablation compared with radiofrequency ablation(contact force), in the treatment of persistent AF.

DETAILED DESCRIPTION:
The hypotheses for this study is that cryothermal energy is as effective and safe as using radiofrequency energy in the treatment of persistent AF and is associated with a better long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* persistent Atrial Fibrillation; Intolerant to antiarrhythmic medication; Both male or female; Age from 18 to 75 years old.

Exclusion Criteria:

* Acute myocardial infarction; Coronary artery stent history; Acute severe stroke; Abnormal liver and renal function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful Pulmonary Vein Isolation | in one year

CONTACTS AND LOCATIONS:
Overall Officials: Baopeng Tang, Study Chair — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China